CLINICAL TRIAL: NCT02133092
Title: Prospective Study in Belgian Children Hospitalized With Respiratory Syncytial Virus Related Acute Respiratory Infections
Brief Title: A Study in Belgian Children Hospitalized With Respiratory Syncytial Virus Related Acute Respiratory Infections
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR103179; ObserveRSV0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Respiratory Syncytial Virus
Keywords: Respiratory syncytial virus; RSV; Lower respiratory tract infection; LRTI; Acute respiratory infection; Belgian children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with respiratory syncytial virus (RSV) infection: The RSV infection is laboratory confirmed
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study. The children hospitalized with lower respiratory tract infection (LRTI) with a laboratory confirmed RSV infection will be monitored for maximum 7 days or until hospital discharge.

SUMMARY:
The purpose of the study is to assess viral kinetics and clinical symptoms kinetics in pediatric patients hospitalized with Respiratory Syncytial Virus (RSV) confirmed lower respiratory tract infection (LRTI).

DETAILED DESCRIPTION:
This is an exploratory prospective study (a study in which the patients are identified and then followed forward in time for the outcome of the study). The study will consist of two phases: a screening phase (Day 1) and an assessment phase (Day 2 to Day 7). During screening phase, in pediatric patients hospitalized with LRTI and from whom the informed consent form was obtained, diagnosis of RSV infection will be performed within 24h from the hospital admission, using a SOFIA POC test on nasal specimens. During the assessment phase the collection of nasal specimens will be done daily for a maximum of 6 days (Day 2 to Day 7 of hospitalization) or until patient discharge from hospital. Approximately 50 patients will be enrolled in this study. The total duration of the study for each participant will be approximately 7 days. The study duration will extend during 1-3 RSV epidemic seasons, or until the targeted number of 50 RSV hospitalized children have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Legal representative has provided Ethics Committee approved written informed consent prior to any study-related procedure(s) being performed and is willing to allow the participation of child to the study for 7 consecutive days or until hospital discharge (whatever comes first)
* Participant hospitalized with lower respiratory tract infection (LRTI) during respiratory syncytial virus (RSV) epidemics, within 24h of hospitalization. The diagnosis of LRTI will follow the standard medical procedure in the hospital unit
* Onset of acute respiratory symptoms was less than or equal to 5 days ago
* For the participation in the assessment phase the hospitalized participant will have an RSV confirmed infection based on SOFIA RSV point of care (POC) test

Exclusion Criteria:

- Participant does not fulfill the inclusion criteria

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients hospitalized with a laboratory confirmed Respiratory Syncytial Virus (RSV) lower respiratory tract infection.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Rate of Respiratory Syncytial Virus (RSV) Viral Clearance | Day 1 to Day 3
  RSV viral clearance, defined as the change in log viral load (VL) from Day 1 to Day 3, where the VL is measured in nasal specimens with quantitative reverse transcript poly cycle reaction (qRT-PCR).

SECONDARY OUTCOMES:
Change From Baseline in Clinical Symptoms Score (CSS) | Day 1 (baseline) to Day 3
  The severity of the RSV disease will be assessed using CSS. CSS will be computed based on clinical parameters (O2 saturation, heart rate, respiratory rate) and lung auscultation examination. CSS score ranges from 0 (best) to 15 (worst). Higher scores indicate worsening.
Change From Baseline in Medical Support Score (MSS) | Day 1 (baseline) to Day 3
  The severity of the RSV disease will be assessed using MSS. MSS will take into account the use of supplementary oxygen, the request for mechanical ventilation, intensive care unit admission and the length of hospitalization. The MSS score ranges from 0 (best) to 5 (worst). Higher scores indicate worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- Belgium (4):
  - Bruges
  - Leuven
  - Lier
  - Ostend

REFERENCES:
- [Derived] Proesmans M, Rector A, Keyaerts E, Vandendijck Y, Vermeulen F, Sauer K, Reynders M, Verschelde A, Laffut W, Garmyn K, Fleischhackl R, Bollekens J, Ispas G. Risk factors for disease severity and increased medical resource utilization in respiratory syncytial virus (+) hospitalized children: A descriptive study conducted in four Belgian hospitals. PLoS One. 2022 Jun 6;17(6):e0268532. doi: 10.1371/journal.pone.0268532. eCollection 2022. PMID 35666728